CLINICAL TRIAL: NCT07401758
Title: Clinical Eficacy of Extracorporeal Shock Wave Therapy on Patellar Tendon Combined With Center of Coordination Point in the Fascial Manipulation for Patellar Tendinitis:A Randomized Controlled Trial.
Brief Title: Clinical Eficacy of Extracorporeal Shock Wave Therapy on Patellar Tendinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2025-946-02
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Shock Wave Threapy for Patellar Tendinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Extracorporeal shockwave therapy was performed not only on the patellar tendon but also at the coordination centre points marked after assessment by a fascia therapist .
  Interventions: Procedure: Extracorporeal Shock Wave Therapy on Patellar Tendon Combined with Center of Coordination Point
- Control Group (Active Comparator): Extracorporeal shockwave therapy was performed only on the patellar tendon .
  Interventions: Procedure: Extracorporeal Shock Wave Therapy only on Patellar Tendon

INTERVENTIONS:
Procedure: Extracorporeal Shock Wave Therapy on Patellar Tendon Combined with Center of Coordination Point — Extracorporeal shockwave therapy was performed on the patellar tendon (Belgium Gymna Shock Master 500 Extracorporeal Shockwave Therapy Device) with a frequency of 8Hz and energy of 2.0Bar, for a total of 2000 shocks; shockwave therapy was performed at the coordination centre points marked after assessment by a fascia therapist (Belgium Gymna Shock Master 500 Extracorporeal Shockwave Therapy Device) with a frequency of 8Hz and energy of 2.0Bar, for a total of 4000 shocks. The patient underwent a total of 3 treatment courses, with an interval of 1 week between each course.
  Arms: Experimental Group
Procedure: Extracorporeal Shock Wave Therapy only on Patellar Tendon — Extracorporeal shockwave therapy was performed only on the patellar tendon (Belgium Gymna Shock Master 500 Extracorporeal Shockwave Therapy Device) with a frequency of 8Hz and energy of 2.0Bar, for a total of 6000 shocks.The patient underwent a total of 3 treatment courses, with an interval of 1 week between each course.
  Arms: Control Group

SUMMARY:
This study is a randomized controlled trial. Patients diagnosed with patellar tendinitis and meeting the criteria for shockwave therapy were included. Relevant clinical data and assessments were collected upon enrollment and after obtaining informed consent. Randomization was performed using a random number table: the experimental and control groups. Based on the group assignments, the experimental group received either patellar tendon combined with fascial therapy coordinated centre point shock wave treatment, while the control group received only shockwave therapy for the patellar tendon. The treatments were performed by a rehabilitation therapist with extensive clinical experience. Data on participant pain and knee joint function were collected using the Visual Analogue Scale (VAS) and the Lysholm Knee Scoring System at baseline and on the day following completion of all treatments. Data on the thickness of the patellar tendon on the affected side of the knee were collected using a portable musculoskeletal ultrasound imaging system. Follow-up assessments and data collection on pain and knee joint function were conducted using the VAS and Lysholm Knee Scoring Scale one month and three months after the completion of all treatments to compare changes before and after treatment and to evaluate whether patellar tendon combined with fascial therapy coordinated centre point shock wave therapy has superior short-term and medium-term maintenance efficacy for patellar tendinitis compared with simple patellar tendon shock wave therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 45 yearsWillingness to sign an informed consent form and ability to cooperate with the treatment and follow-up aspects of this study.
2. Meeting the diagnostic criteria for patellar tendinitis as outlined in "Practical Sports Medicine" (2023 edition)
3. Knee joint pain with a VAS score of ≥3 and ≤7
4. No other orthopedic or neurological conditions that could affect lower limb strength or mobility
5. Willingness to sign an informed consent form and ability to cooperate with the treatment and follow-up aspects of this study

Exclusion Criteria:

1. History of knee joint surgery within the past year
2. Presence of knee pain due to other causes, or conditions that affect the knee joint or impact its function (including but not limited to: transient synovitis, bone tuberculosis, bone tumors, acute traumatic arthritis, suppurative arthritis, rheumatoid arthritis, metabolic bone diseases, psoriatic arthritis, gouty arthritis, bone necrosis, ankylosing spondylitis, or active infections)
3. Presence of chronic knee pain caused by other reasons (such as post-herpetic neuralgia, osteoporosis, etc.)
4. Contraindications for shockwave therapy, such as deep venous thrombosis in the lower extremities, bleeding disorders or coagulation dysfunction, pregnancy, cognitive dysfunction, etc.
5. Presence of cancerous tumors, severe bronchiectasis, acute suppurative inflammation, high fever, active pulmonary tuberculosis, heart failure, severe anemia, cerebrovascular diseases, or the presence of a cardiac pacemaker implanted in the body
6. Inability to participate in the trial due to other health issues, such as sudden severe trauma, sudden severe infectious diseases, etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the change in pain intensity over a follow-up period of 3 months after treatment | Baseline and Day 105
  Determine the medium-term maintenance effect of pain relief before and after treatment. Use the Visual Analogue Scale (VAS) to quantitatively assess changes in pain intensity at the 3-month follow-up after treatment. At baseline and at 3 months after the completion of all treatments, the assessment is carried out using the Visual Analogue Scale by a trained therapist who is not involved in the intervention treatment or data analysis.

SECONDARY OUTCOMES:
The changes in pain intensity measured both on the day following treatment and during the follow-up period of one month | Baseline, Day 15 and Day 45
  Determine the early changes in the intensity of knee pain in patients: assessed at baseline, on the day all treatments were completed, and one month after all treatments were completed, using a visual analogue scale by a trained therapist not involved in the intervention treatment or data analysis.
the changes in the Lysholm knee scoring scale after treatment, as well as during follow-up visits after one and three months. | Baseline, Day 15, Day 45 and Day 105
  Changes in patient knee joint function: At baseline, on the day of completion of all treatments, and at 1 and 3 months after completion of all treatments, the function of the patient's affected knee joint was assessed by a trained therapist not involved in the intervention treatment or data analysis using the Lysholm Knee Scoring Scale.
the change in the thickness of the patellar tendon on the day following treatment | Baseline and Day 15
  Changes in the thickness of the patient's knee patellar tendon: At baseline and on the day after all treatments were completed, the thickness of the patellar tendon of the affected knee was assessed using a portable musculoskeletal ultrasound imaging system by a trained therapist who did not participate in the intervention treatment or data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- 中山大学孙逸仙纪念医院, Guangzhou, Guangdong, China

DOCUMENTS (2):
  • Study Protocol (2025-12-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT07401758/Prot_000.pdf
  • Informed Consent Form (2025-11-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT07401758/ICF_001.pdf